CLINICAL TRIAL: NCT04672902
Title: Single-operator Cholangioscopy and Electrohydraulic Lithotripsy for the Treatment of Mirizzi Syndrome: A Case Series
Brief Title: Treatment of Mirizzi Syndrome
Status: Completed | Type: Observational
Sponsor: Tecnologico de Monterrey (Other)
Responsible Party: Sponsor
Other Study IDs: MS2012
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Mirizzi Syndrome; Cholelithiasis; Acute Cholecystitis
MeSH Terms: conditions — Mirizzi Syndrome; Cholelithiasis; Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Single-operator cholangioscopy guided electrohydraulic lithotripsy — Single-operator cholangioscopy guided electrohydraulic lithotripsy has the advantage of providing direct visualization of the bile ducts, enabling a single physician to diagnose and perform the therapeutic intervention in a single procedure.

SUMMARY:
Mirizzi syndrome is an infrequent complication of long-standing cholelithiasis. Extrinsic compression of the common hepatic duct is usually caused by an impacted stone in Hartmann's pouch or cystic duct resulting in the development of cholecystobiliary fistula. This syndrome is classified based on the presence and severity of cholecystobiliary fistula. Mirizzi syndrome is challenging to diagnose preoperatively and may require complex biliary surgical procedures for resolution. Endoscopic treatment is a safe alternative with a high success rate. Single-operator cholangioscopy combined with lithotripsy has been shown to have a 90-100% success rate in the treatment of biliary stones. Herein, A single center experience treating Mirizzi syndrome with single-operator cholangioscopy guided electrohydraulic lithotripsy is presented. Difficult management of Mirizzi syndrome has led to research of new treatment options to minimize the risk of high rate complications. Single-operator cholangioscopy in combination with laser lithotripsy is an adequate and safe alternative for the treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients with a preoperative diagnosis of Mirizzi Syndrome
* Patients with a common bile duct dilatation

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with an inconclusive biliary diagnosis
* Patients without a diagnosis of Mirrizi Syndrome
* Patients without common bile duct dilatation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A 34-year-old female, A 54-year-old male, A 40-year-old female. with diagnosed Mirizzi Syndrome by an image study, with a concomitant common bile duct dilatation.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Resolution of the common bile duct compression by an extrinsic gallbladder stone, with minimally invasive procedure such as single operator cholangioscopy, combined with lithotripsy | 2019-2020
  Single operator cholangioscopy, combined with lithotripsy, will be use for treating patients with Mirizzi syndrome, while avoiding open surgery, and subsequent lesions to the biliary ducts. Post surgical morbidity will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela Nacional de Medicina, Tecnologico de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided